CLINICAL TRIAL: NCT03269604
Title: Effectiveness of Three Different Times of Starting Antibiotic Prophylaxis in Patients With Asymptomatic Bacteriuria Scheduled for Urological Surgery. A Randomized Multicentric Clinical Trial
Brief Title: Effectiveness of Three Times of Starting Antibiotic Prophylaxis in Patients With Asymptomatic Bacteriuria.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jorge Andres Ramos Castaneda (Other)
Responsible Party: Sponsor-Investigator, Jorge Andres Ramos Castaneda, Ph. D. student in Public Health, CES University
Organization: CES University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1075237598
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Asymptomatic Bacteriuria; Antibiotic Prophylaxis
Keywords: Urological Surgery; Bacterial resistance
MeSH Terms: interventions — Chemoprevention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: A single blinding will be performed. To the database will be categorized the variable "duration of prophylaxis" so that the person in charge of analysing the data, does not know the true allocation of each of the participants. At the end of the tabulation and analysis of the data, the true allocation will be known.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prophylactic antibiotic five days previous to the procedure (Active Comparator): Prophylactic antibiotic during five days previous to the procedure.
  Interventions: Procedure: Prophylactic antibiotic during five days previous to the procedure
- Prophylactic antibiotic three days previous to the procedure (Active Comparator): Prophylactic antibiotic during three days previous to the procedure.
  Interventions: Procedure: Prophylactic antibiotic during three days previous to the procedure
- Only a single dose of Prophylactic antibiotic (Experimental): Only a single dose of Prophylactic antibiotic on the day of the procedure
  Interventions: Procedure: Only a single dose of Prophylactic antibiotic

INTERVENTIONS:
Procedure: Prophylactic antibiotic during five days previous to the procedure — Prophylactic antibiotic during five days previous to the procedure.
  Arms: Prophylactic antibiotic five days previous to the procedure
Procedure: Prophylactic antibiotic during three days previous to the procedure — Prophylactic antibiotic during three days previous to the procedure.
  Arms: Prophylactic antibiotic three days previous to the procedure
Procedure: Only a single dose of Prophylactic antibiotic — This group will receive a single dose of antibiotic 90 ± 20 minutes prior to the start of the surgical procedure (incision)
  Arms: Only a single dose of Prophylactic antibiotic

SUMMARY:
Asymptomatic bacteriuria (AB) is the isolation of a bacterium in a sample of urine appropriately collected from a person who does not have signs or symptoms of urinary infection. It is common in diabetic women, in pregnant women, in men over 60 years and in patients with spinal cord injury.

There is clinical evidence that AB should be treated in patients who will be operated on with urologic surgery because of the risk of presenting infectious complications; however, the timing of initiating antibiotic therapy has not been established, even in some studies the prophylaxis has been considered from one to seven days prior to the procedure, without determining the differences in the outcome for each one of the interventions and causing an undue and risky use of antibiotics.

A randomized, parallel-design, single-masked clinical trial will be performed to compare and analysis the bloodstream infections, surgical site infections, readmissions and hospital stay in three intervention groups, 1) those receiving antibiotics during the previous 5 days to the procedure; 2) 3 days prior to the procedure; and 3) those who receive only a single dose of antibiotic on the day of the procedure.

The main expected result is to identify the timing of initiation of antibiotic prophylaxis in urological procedures in patients with asymptomatic bacteriuria, with the purpose of diminishing the bloodstream and of the surgical site infections. If it is scientifically demonstrated that those patients who receive a single dose of antibiotic on the same day of the procedure, have the same safety and effectiveness compared to the other two groups, would reduce hospital stay, surgical waiting time and indiscriminate use of antibiotics that generate multidrug-resistant microorganisms, thus generating an impact on Public Health and on the quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with asymptomatic bacteriuria identified with a urine culture prior to the surgical procedure and with a microorganism that meets the following criteria: 1) gram-negative bacteria in the enterobacterial family and non-fermenting bacilli; 2) Bacteria with resistance profile has a therapeutic option that reaches therapeutic concentration in urine.
* Patients scheduled for urological procedures, such as: transurethral resection of the prostate, open prostatectomy, cystoscopy, extracorporeal lithotripsy and flexible ureterorenoscopy.
* Informed consent

Exclusion Criteria:

* Patients with chronic renal failure; with immunosuppressive status secondary to glucocorticoid consumption, haematological or solid organ neoplasms undergoing chemotherapy or radiation therapy or neutropenia.
* Patients with active infection or clinical criteria of urinary infection.
* Patients who voluntarily do not want to participate in the study.
* Patients who can not give informed consent under reasonable or vulnerable conditions.
* Patients who present type I allergy to penicillin.
* Patients who have scheduled surgeries combined with a discipline different to urology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Bloodstream infection | 30 days
  An infectious process characterized by the presence of some bacteria in the bloodstream. The patient should have one or more positive blood cultures, where the cultured organism is not related to an infection elsewhere, and has signs of infection, such as fever, hypotension or tachycardia.

SECONDARY OUTCOMES:
Surgical Site Infection: | 30 days
  It can occur up to 30 days (or a year when a prosthetic component is involved) of a surgical procedure in some part of the body where it was manipulated in surgery. The SSI is classified as superficial, deep or organ space, depending on the type of tissue involved.
Length of hospital stay | 30 days
  Difference in days between the date of discharge and of the surgical procedure.
Re-entry to hospitalization | 30 days
  Re hospitalization after the surgical procedure due to SSI or bloodstream.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad CES, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Undecided